CLINICAL TRIAL: NCT00380822
Title: Double-Blind Study of Miglitol in Japanese With type2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanwa Kagaku Kenkyusho Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MG1001
Record Dates: First submitted 2006-09-25; First posted 2006-09-27 (Estimated); Last update posted 2006-09-27 (Estimated); Status verified 2006-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: alpa-glucosidase inhibitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — miglitol

INTERVENTIONS:
Drug: miglitol

SUMMARY:
To investigate the efficacy and safety of miglitol in Japanese patients with type 2 diabetes that is insufficiently controlled diet alone.

ELIGIBILITY:
Inclusion Criteria:

* Type2 diabetic patient on Dietary Therapy
* Criteria for postprandial plasma glucose and HbA1c are met

Exclusion Criteria:

* Type1 diabetes
* Patients treated with antidiabetic drugs or Insulin

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Clinical study Group, Clinical Development Dept., Study Director — Sanwa Kagaku Kenkyusho Co., Ltd.
Locations (27):
- Japan (27):
  - Aichi
  - Chiba
  - Fukuoka
  - Gunma
  - Hiroshima
  - Hyōgo
  - Ibaraki
  - Ishikawa
  - Kumamoto
  - Kyoto
  - Mie
  - Miyagi
  - Nagasaki
  - Niigata
  - Numakunai
  - Okayama
  - Osaka
  - Ōita
  - Saga
  - Saitama
  - Shiga
  - Shimane
  - Shizuoka
  - Tokyo
  - Toyama
  - Yamagata
  - Yamaguchi